CLINICAL TRIAL: NCT01349114
Title: Effect of the Direct Renin Inhibitor Aliskiren on Endothelial Function and Arterial Stiffness in Diabetic Subjects
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor requested termination.
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, David Calhoun, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: F110124007
Record Dates: First submitted 2011-05-04; First posted 2011-05-06 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-04

CONDITIONS: Diabetes; Pre-hypertension; Hypertension
Keywords: aliskiren; endothelial function; hypertension
MeSH Terms: conditions — Diabetes Mellitus; Prehypertension; Hypertension | interventions — aliskiren; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- aliskiren 300 mg once daily for 12 weeks (Active Comparator): aliskiren 300 mg daily
  Interventions: Drug: aliskiren 300 mg once daily
- Sugar pill/ placebo (Placebo Comparator): Patients were double-blind placebo-controlled randomized to either aliskiren 300 mg once daily or sugar pill/ placebo
  Interventions: Drug: Placebo/sugar pill

INTERVENTIONS:
Drug: aliskiren 300 mg once daily — aliskiren 300 mg daily
  Other Names: Tekturna
  Arms: aliskiren 300 mg once daily for 12 weeks
Drug: Placebo/sugar pill — Sugar pill/placebo
  Arms: Sugar pill/ placebo

SUMMARY:
The study will evaluate the effects of the direct renin inhibitor, aliskiren, on flow-mediated dilation of the brachial artery and on central aortic pressure in diabetic patients with pre-hypertension or Stage 1 hypertension.

DETAILED DESCRIPTION:
Patients are double-blind placebo-controlled randomized to either aliskiren or sugar pill/placebo. Effects on blood parameters and arteries are evaluated in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* prehypertension or Stage 1 hypertension

Exclusion Criteria:

* Type 1 diabetes
* Stage 2 hypertension
* CKD
* recent MI, revascularization, CVA or TIA

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Calhoun, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Aliskiren: aliskiren 300 mg daily
- Sugar Pill/Placebo: Sugar pill/placebo arm
Period: Overall Study
Arm/Group | Aliskiren | Sugar Pill/Placebo
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Sugar pill/placebo
- Total: Total of all reporting groups
Arm/Group | Aliskiren | Placebo | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (11) | 63.4 (8.3) | 60.7 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Flow-mediated Dilation
Description: Flow-mediated dilation of the brachial artery assessed by ultrasound to evaluate improvement of arterial functioning by % of dilation after non-invasive occlusion
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: percentage of flow-mediated dilation
Groups:
- Placebo: Sugar pill/ placebo
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 10 | 11
percentage of flow-mediated dilation | 7.9 (2.5) | 4.1 (1.3)

2. Secondary Outcome: Mean Central Aortic Pressure at 3 Months
Description: Baseline to 3 months after Aliskiren/PLC, reported value at 3 months after start of study of central aortic pressure assessed by non-invasive applanation tonometry ( SphygmoCor, Atcor)
Time Frame: 3 months after start of study
Population: Aortic pressure indicates the augmentation pressure (AP) in mmHg derived from the radial artery waveform.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Aliskiren: aliskiren 300 mg daily
  aliskiren: aliskiren 300 mg daily
- Placebo: placebo: placebo
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 10 | 11
mm Hg
  aortic systolic blood pressure | 113.4 (12.0) | 122.3 (9.6)
  aortic diastolic blood pressure | 78.9 (8.9) | 83.3 (9.9)
  aortic pressure | 7.1 (7.2) | 10.3 (5.7)

ADVERSE EVENTS:
Arm/Group | Aliskiren | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11

LIMITATIONS AND CAVEATS:
Early termination leading to smaller number of subjects analyzed then anticipated, no adverse effects within the aliskiren group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No